CLINICAL TRIAL: NCT04265690
Title: A Multi-Component Nutrition Program for Pregnant and Parenting Teens, a Pilot Study
Brief Title: A Multi-Component Nutrition Program for Pregnant and Parenting Teens
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study never launched due to several COVID-19 related barriers.
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H-39461
Record Dates: First submitted 2020-02-09; First posted 2020-02-11 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Adolescent Behavior; Pregnancy Related; Postpartum
Keywords: Healthy eating behaviors; Eating competence; Centering pregnancy; Centering parenting
MeSH Terms: conditions — Adolescent Behavior

STUDY DESIGN:
Intervention Model Description: For this proof of concept/pilot trial, we will assess the feasibility and impact of this multi-component nutrition program on improving healthy eating behaviors and eating competence. However, because we are proposing a proof of concept pilot and feasibility study, in our experience and that of others, our proposed sample size generally provides sufficient data to estimate subject retention, distribution of variables and feasibility as we plan for a larger-multi-site RCT of the proposed study. We expect our intervention to demonstrate the feasibility of the intervention in a clinic setting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Teen and Tot Centering subjects (Experimental): The cooking classes and text messages will supplement the subject's standard of care by incorporating text messages and a cooking class.
  Interventions: Behavioral: Cooking classes; Behavioral: Text messages

INTERVENTIONS:
Behavioral: Cooking classes — Participants will receive 2 cooking classes (each 1-hour long) during their Centering group-care visit at the BMC teaching kitchen, taught by a Registered Dietitian. The recipes taught during the cooking classes will follow the Special Supplemental Nutrition Program for Women, Infants, and Children, the 2015-2020 Dietary Guidelines for Americans, and recommendations from The American College of Obstetricians and Gynecologists.
Behavioral: Text messages — Participants will receive text messages, through a password secured phone, based on their content and frequency preferences.

SUMMARY:
Improving nutrition during pregnancy is critical for maternal and child health, but even more so among pregnant adolescents. Several studies have shown that poor nutrition and diet quality during pregnancy is related to adverse health outcomes among both the mother and the infant. During pregnancy, the fetus's nutrition and diet quality is largely dependent on the mother. A teenage mother is in a vulnerable position because she needs to meet the demands of her own growth and development in addition to the growth and development of her baby, which can be extremely challenging, especially for mothers who are from disadvantaged communities. Surprisingly, given their unique needs, there is limited literature on multicomponent behavioral interventions that adequately address the unique nutritional needs of pregnant adolescent women and their fetuses, which is why interventions targeted at promoting healthy behaviors among low-income, racially diverse pregnant teens should be a public health priority, particularly in the U.S. This study aims to assess whether a multicomponent behavioral intervention improves intention, initiation, and sustained healthy eating behaviors and eating competence among Pregnant adolescents (second trimester) and Postpartum adolescent mothers (<6 months).

ELIGIBILITY:
Inclusion Criteria:

* 15-23 years of age
* be at least 3 months pregnant; or
* have a baby less than 2 years old
* be participating in Teen and Tot Centering group-care visits

Exclusion Criteria:

* None

Ages: 15 Years to 23 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Change in eating competence | Baseline, 3 months
  Eating competence will be measured using the ecSatter Inventory (EcSI 2.0) which assesses: eating attitudes, food acceptance, food regulation, and contextual skills. The 16 item EcSI 2.0 questionnaire uses a 5-point likert scale with scores from 3 to 0 [Always=3; Often =2; Sometimes=1, Rarely=0; Never=0]. Total EcSI 2.0 scores range from 0 to 48. Higher EcSI 2.0 scores are correlated with better eating competence. Eating competence cutoff is 32 and above.

SECONDARY OUTCOMES:
Change in nutrition knowledge | Baseline, 3 months
  Assess nutrition knowledge based on the General Nutrition Knowledge Questionnaire (GNKQ). The scale assesses: dietary recommendations, food groups, healthy food choices, and diet, disease, and weight associations. The GNKQ questionnaire is 88 items. The highest total GNKQ score is 88 and the lowest is 0. Higher GNKQ scores are correlated with better nutrition knowledge.
Cooking class acceptability | 3 months
  The acceptability of the cooking classes will be assessed by a short survey with 4 questions and a 5-point likert scale that was made by the investigator. The survey will ask about their opinions about the cooking classes' nutrition information delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Marisol De Ornelas, Principal Investigator — Boston Medical Center

IPD SHARING:
Plan to Share IPD: No